CLINICAL TRIAL: NCT05989074
Title: All Women A Multicenter Randomized Clinical Trial Comparing Self-expanding ALLEGRA Valve to Any Other Balloon-expandable Valve in a Women Population
Brief Title: All Women Comparing Self-expanding ALLEGRA Valve to Any Other Balloon-expandable Valve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ceric Sàrl (Industry)
Collaborators: Biosensors International (Other); European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BSR-14
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-08

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALLEGRA (Experimental): ALLEGRA Delivery System TF will be administered.Patient will receive Anticoagulation medication according to the site-specific standard of care
  Interventions: Device: ALLEGRA TAVI System TF
- Balloon-expandable TAVI (Active Comparator): Patient will receive any kind of CE-marked balloon-expandable valve, and anticoagulation medication according to the site-specific standard of care
  Interventions: Device: Ballon-expandable valve system

INTERVENTIONS:
Device: ALLEGRA TAVI System TF — Patients receive ALLEGRA TAVI System TF. Patient will receive medication according to routine practice of the hospital
  Arms: ALLEGRA
Device: Ballon-expandable valve system — Patients receive any kind of CE-marked balloon expandable valve system, used at the hospital. Patient will receive medication according to routine practice of the hospital.
  Arms: Balloon-expandable TAVI

SUMMARY:
Study is aimed to demonstrate that the self-expandable Allegra TAVI system provides lower mean gradient assessed by TTE compared to balloon-expandable valve systems in a female patient population with symptomatic severe aortic stenosis

DETAILED DESCRIPTION:
Study is aimed to demonstrate that the self-expandable Allegra transcatheter aortic valve implantation (TAVI) system provides lower mean gradient assessed by Transthoracic Echo (TTE) at 30 days post procedure, compared to balloon-expandable valve systems in a female patient population with symptomatic severe aortic stenosis.

Patients in both arm will receive anticoagulants according to routine practice of the hospital.

Patients will be followed-up until 1 year after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex
2. Age ≥ 75 years (according to ESC/EACTS, Guidelines for the management of valvular heart disease)
3. Severe calcific aortic valve stenosis defined as follows: high-gradient aortic stenosis (mean pressure gradient across aortic valve > 40 mmHg or peak velocity > 4.0 m/s) Symptomatic aortic valve stenosis with New York Heart Association (NYHA) Class ≥II
4. ECG-gated Multi-Slice Computed Tomographic (MSCT) measurements determined an aortic annulus perimeter-derived average diameter >19 mm and <27.4 mm or area-derived diameter >18 and <28 mm
5. Anatomy suitable for trans-femoral TAVI for both devices used in the study, including a minimum femoral diameter of 6 mm.
6. Subject with a documented local Heart Team (HT) indication for TF TAVI
7. Life expectancy longer than 1 year.
8. Willingness to undergo clinical and echocardiographic follow-up after the procedure.
9. Subject can understand the purpose of the clinical investigation, has signed voluntarily the informed consent form and is agreeing to the scheduled follow-up requirements

Exclusion Criteria:

1. Male sex
2. Non-calcific acquired aortic stenosis
3. Native unicuspid/bicuspid aortic valve or congenital aortic abnormality
4. Previous implantation of heart valve in any position
5. Severe aortic regurgitation (> 3+)
6. Severe mitral regurgitation (> 3+)
7. Severe tricuspid regurgitation (> 3+)
8. Severe left ventricular dysfunction (Left Ventricular Ejection Fraction (LVEF) < 30%)
9. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
10. Untreated cardiac conduction disease in need of pacemaker implantation
11. Evidence of acute Myocardial Infarction (MI) less than 30 days before signing informed consent
12. Any need for emergency surgery
13. Any active bleeding that precludes anticoagulation
14. Liver failure (Child-C)
15. End-stage renal disease requiring chronic dialysis or creatinine clearance < 30cc/min
16. Pulmonary hypertension (systolic pressure > 80mmHg)
17. A known hypersensitivity or contraindication to all anticoagulation/antiplatelet regimens (or inability to be anticoagulated for the index procedure), to cobalt chromium, to bovine and/or collagen, glutaraldehyde or contrast media
18. Any medical, social or psychological condition that in the opinion of the investigator precludes the subject from giving appropriate consent or adherence to the required follow-up procedures
19. Currently participating in another drug or device trial (excluding observational registries) for which the primary endpoint has not been assessed
20. Subject under judicial protection, tutorship or curatorship (for France only)

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Biological gender
Enrollment: 130 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Trans-aortic mean gradient measured by TTE 30 days after the TAVI procedure. | At 30 Days
  Trans-aortic mean gradient measured by TTE 30 days after the TAVI procedure.

SECONDARY OUTCOMES:
Technical success assessed by composite criteria | Up to the end of the time when patient exit the procedure room
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Device success assessed by composite criteria | At 30 days
  Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve‡ (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥ 0.25, and less than moderate aortic regurgitation)
Early safety assessed by composite criteria | At 30 days
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from Valve Academic Research Consortium (VARC) type 2-4 bleeding (in trials where control group is surgery, it is appropriate to include only Type 3 and 4 bleeding)
  * Freedom from major vascular, access-related, or cardiac structural complication
  * Freedom from acute kidney injury stage 3 or 4
  * Freedom from moderate or severe aortic regurgitation
  * Freedom from new permanent pacemaker due to procedure-related conduction abnormalities
  * Freedom from surgery or intervention related to the device
Clinical efficacy assessed by composite criteria | At 1 year
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from hospitalization for procedure- or valve-related causes
  * Freedom from Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score <45 or decline from baseline of >10 point (i.e. Unfavourable Outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Alaide Chieffo, Prof, Principal Investigator — Ospedale San Raffaele; Ignacio Cruz-Gonzalez, Prof, Principal Investigator — University of Salamanca

IPD SHARING:
Plan to Share IPD: Undecided